CLINICAL TRIAL: NCT06466213
Title: Acute Effects of Three Different Types Single Leg Exercise in Copd
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Kocaaga, principal investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GO23-193
Record Dates: First submitted 2024-05-17; First posted 2024-06-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single session one leg exercise intervantion in COPD (Experimental): first session: single session leg Continuous exercise intervantion will be applied to COPD. Unilaterally single leg continuous exercise will be performed as only one session
  second session : single session leg high intensity interval exercise intervantion will be applied to COPD. Unilaterally single leg hııt exercise will be performed as only one session
  third sessionsingle session leg resistance exercise intervantion will be applied to COPD. Respirocally leg strength (knee extantion ) exercise will be performed
  Interventions: Other: single exercise bout about one-leg exercise

INTERVENTIONS:
Other: single exercise bout about one-leg exercise — cycle exercise includes single leg

SUMMARY:
COPD presents not only respiratory symtoms but also vascular or muscle dysfunction. Exercise training is important for aerobic performance increasing. Generally results show exercise training with both lower limb. Increaed arterial stiffness and muscle oxygenation are observed in COPD. One leg exercise result is not enough to highlight these parameters.

DETAILED DESCRIPTION:
Acute Effects of Three Different Types Single Leg Exercise in Copd

single bout high intensity interval training

single bout continuous exercise training single bout resistance training

ELIGIBILITY:
Inclusion Criteria:

* COPD patients that applied to physiotherapy
* cooperate to test
* no severe ortopedical and neurological disease no severe cardiovascular disease volunteer to study

Exclusion Criteria:

* have an acute exacerbation
* hypoxemia [PaO2] <55 mmHg
* no cooperated to test no volunteer to study having ortophedical and neurological diesase that affecting of tests having severe cardiovascular disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
six minute walk test | beginning, day 1
  six minute walk test in meter

SECONDARY OUTCOMES:
cardiopulmonary exercise test | beginning, day 2
  VO2 max will be recorded as ml/kg/min will be recorded from incremental cycle cpet test
single leg extremity test | beginning, day 3
  VO2 max will be recorded as ml/kg/min will be recorded from incremental cycle cpet test
lung function | beginning, day 1
  FVC in % , FEV1 in %, FEV1/FVC ratio, PEF in % and FEF 25-75 in %
muscle strength (isometric) | beginning day 1
  quadriceps isometric muscle strength will be recorded as kilogram
muscle strength (10 repeated max) | beginning, day 1
  quadriceps 10 repeated max muscle strength will be recorded as kilogram
continous exercise acute (single leg) | beginning day 4
  VO2 max will be recorded as ml/kg/min will be performed from incremental cycle exercise at single session
high intensity interval training acute exercise (single leg) | beginning day 5
  VO2 max will be recorded as ml/kg/min will be performed from incremental cycle exercise at single session
strength training acute exercise (single leg) | beginning day 4,5,6
  VO2 max will be recorded as ml/kg/min will be performed from incremental cycle exercise at single session
muscle oxygenation | beginning day 4,5,6
  minumum muscle oxygenation level will be presented as percentage
arterial stifness | beginning day 2,3, 4,5,6
  Aıx@75 in %

CONTACTS AND LOCATIONS:
Overall Officials: elif kocaaga, ms, Principal Investigator — Hacettepe University
Locations (1):
- Elif Kocaaga, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Evans RA, Dolmage TE, Mangovski-Alzamora S, Romano J, O'Brien L, Brooks D, Goldstein RS. One-Legged Cycle Training for Chronic Obstructive Pulmonary Disease. A Pragmatic Study of Implementation to Pulmonary Rehabilitation. Ann Am Thorac Soc. 2015 Oct;12(10):1490-7. doi: 10.1513/AnnalsATS.201504-231OC. PMID 26291542